CLINICAL TRIAL: NCT01228734
Title: An Open-label, Randomized, Controlled, Multicenter Phase III Trial to Compare Cetuximab in Combination With FOLFOX-4 Versus FOLFOX-4 Alone in the First Line Treatment of Metastatic Colorectal Cancer in Chinese Subjects With RAS Wild-type Status
Brief Title: A Trial to Compare Oxaliplatin, Folinic Acid (FA) and 5-Fluorouracil (5FU) Combination Chemotherapy (FOLFOX-4) With or Without Cetuximab in the 1st Line Treatment of Metastatic Colorectal Cancer (mCRC) in Chinese Rat Sarcoma Viral Oncogene Homolog (RAS) Wild-type Patients
Acronym: TAILOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR62202-057
Record Dates: First submitted 2010-09-09; First posted 2010-10-26 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; RAS wild type; Cetuximab; First line treatment; First occurrence of metastatic colorectal cancer in Chinese subjects with RAS wildtype; status
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab + FOLFOX-4 (Experimental): Subjects received cetuximab in combination with FOLFOX-4 chemotherapy regimen. FOLFOX-4 chemotherapy regimen consists of a combination of oxaliplatin with 5-fluorouracil (5-FU)/folinic acid (FA). Cetuximab was always administered every 7 days with an initial dose of 400 milligram per square meter (mg/m^2) at 5 milligram per minute (mg/min) and 250 mg/m^2 at 10 mg/min for subsequent infusions, followed by oxaliplatin 85 mg/m^2 infused over 120 minutes at least 1 hour later. Following completion of the oxaliplatin infusion or simultaneously with oxaliplatin, FA was administered at a dose of 200 mg/m^2 infused over 120 minutes, on Day 1, Day 2, and every 2 weeks and then 5- FU was administered as a bolus of 400 mg/m^2/day intravenously over 2-4 minutes followed by 600 mg/m^2/day infused over 22 hours, on Day 1, Day 2, and every 2 weeks. All subjects received treatment until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: Cetuximab; Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5Fluorouracil
- FOLFOX-4 (Active Comparator): Subjects received FOLFOX-4 chemotherapy regimen that consists of a combination of oxaliplatin with 5-FU/FA. Oxaliplatin 85 mg/m^2 infused over 120 minutes was administered first or simultaneously with FA at a dose of 200 mg/m^2 infused over 120 minutes on Day 1, Day 2, and every 2 weeks and then 5-FU was administered as a bolus of 400 mg/m^2/day intravenously over 2-4 minutes followed by 600 mg/m^2/day infused over 22 hours on Day 1, Day 2, and every 2 weeks. All subjects received treatment until progression of disease, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5Fluorouracil

INTERVENTIONS:
Drug: Cetuximab — Cetuximab was administered every 7 days at an initial dose of 400 milligram per square meter (mg/m^2) at 5 milligram per minute (mg/min) and 250 mg/m^2 at 10 mg/min for subsequent infusions until progression of disease, withdrawal of consent, or unacceptable toxicity to cetuximab.
  Other Names: Erbitux; C225
  Arms: Cetuximab + FOLFOX-4
Drug: Oxaliplatin — Oxaliplatin 85 mg/m^2 infusion over 120 minutes on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
Drug: Folinic Acid — FA 200 mg/m^2 infusion over 120 minutes on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.
Drug: 5Fluorouracil — 5-FU as a bolus of 400 mg/m^2/day intravenously over 2-4 minutes followed by 600 mg/m^2/day infusion over 22 hours on Day 1, Day 2, and then every 2 weeks until progression of disease, withdrawal of consent, or unacceptable toxicity.

SUMMARY:
The purpose of this study was to assess whether the progression free survival (PFS) time with FOLFOX-4 plus cetuximab is longer than that with FOLFOX-4 alone as first-line treatment for mCRC in Chinese subjects with RAS wild-type tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent (first and second)
* Chinese with Chinese citizenship
* Male or female subjects greater than or equal to (>=) 18 years of age
* Medically accepted effective contraception if procreative potential exists (applicable for both male and female subjects until at least 90 days after the last dose of trial treatment)
* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* First occurrence of metastatic disease (not curatively resectable) RAS wild-type status in tumor tissue
* At least one measurable lesion by computer tomography (CT) or magnetic resonance imaging (MRI) according to RECIST (not in an irradiated area)
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at trial entry
* White blood cell count >= 3 × 10x9/L with neutrophils >= 1.5 × 10x9/L, platelet count >= 100 × 10x9/L and hemoglobin >= 6.21 mmol/L (10 g/dL)
* Total bilirubin <= 1.5 × upper limit of reference range
* Aspartate transaminase (AST) and alanine transaminase (ALT) <= 2.5 × upper limit of reference range or <= 5 × upper reference range in subjects with liver metastasis
* Serum creatinine <= 1.5 × upper limit of reference range
* Recovery from relevant toxicity due to previous treatment before trial entry

Exclusion Criteria:

* Previous chemotherapy for CRC except adjuvant treatment if terminated > 9 months (oxaliplatin-based chemotherapy) or > 6 months (non-oxaliplatin-based chemotherapy) before the start of treatment in this trial
* Radiotherapy or surgery (excluding prior diagnostic biopsy) in the 30 days before trial treatment
* Previous treatment with monoclonal antibody therapy, vascular endothelial growth factor (VEGF) pathway-targeting therapy, epidermal growth factor receptor (EGFR) pathway-targeting therapy, or other signal transduction inhibitors
* History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation
* Renal replacement therapy
* Intake of any investigational medication within 30 days before trial entry
* Concurrent chronic systemic immune therapy or hormone therapy except physiologic replacement
* Granulocyte colony stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF) within 3 weeks of trial entry (these growth factors may be used during the trial thereafter)
* Other non-permitted concomitant anticancer therapies
* Known brain metastasis and/or leptomeningeal disease. Subjects with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis
* Previous malignancy other than CRC in the last 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 5 years, or left ventricular ejection fraction below the institutional range of normal on a baseline multiple gated acquisition scan or echocardiogram
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Active clinically serious infections (> grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0), including active tuberculosis
* Known and declared history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Peripheral neuropathy > grade 1
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
* Uncontrolled diabetes mellitus, pulmonary fibrosis, acute pulmonary disorder, interstitial pneumonia, or liver failure
* Known hypersensitivity or allergic reactions against any of the components of the trial treatments
* Pregnancy (absence to be confirmed by serum β-human chorionic gonadotropin test) or breastfeeding
* Ongoing alcohol or drug abuse
* Presence of a medical or psychological condition that would not permit the subject to complete the trial or sign informed consent
* Participation in another clinical trial within the past 30 days
* Other significant disease that in the investigator's opinion should exclude the subject from the trial
* Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Beijing, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (25):
- China (25):
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - Fuzhou General Hospital, Fuzhou, Fujian
  - First Hospital Affiliated to Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Jilin Cancer Hospital, Changchun, Jilin
  - First Affiliated Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - 307 Hospital of PLA, Beijing
  - The General Hospital of the People's Liberation Army, Beijing
  - Affiliated Hospital of Bengbu Medical College, Bengbu
  - The Xiangya 2nd Hospital of Central South University, Changsha, Hunan
  - Southwest Hospital, Chongqing
  - Yunnan Provincial Tumor Hospital, KunMing, Yunnan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Fudan University Zhongshan Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Shuzhou, Jiangsu
  - Tianjin People's Hospital, Tianjin
  - Xijing Hospital the 4th Military Medical University of PLA, Xi'an

REFERENCES:
- [Derived] Wang H, Huang L, Gao P, Zhu Z, Ye W, Ding H, Fang L. Cost-effectiveness analysis of cetuximab combined with chemotherapy as a first-line treatment for patients with RAS wild-type metastatic colorectal cancer based on the TAILOR trial. BMJ Open. 2020 Feb 12;10(2):e030738. doi: 10.1136/bmjopen-2019-030738. PMID 32051297
- [Derived] Bai L, Zhang P, Zhou K, Liao W, Li Q. Cost-Effectiveness Analysis of First-Line Cetuximab Plus Leucovorin, Fluorouracil, and Oxaliplatin (FOLFOX-4) versus FOLFOX-4 in Patients with RAS Wild-Type Metastatic Colorectal Cancer. Cancer Manag Res. 2019 Dec 12;11:10419-10426. doi: 10.2147/CMAR.S219318. eCollection 2019. PMID 31849531
- [Derived] Qin S, Li J, Wang L, Xu J, Cheng Y, Bai Y, Li W, Xu N, Lin LZ, Wu Q, Li Y, Yang J, Pan H, Ouyang X, Qiu W, Wu K, Xiong J, Dai G, Liang H, Hu C, Zhang J, Tao M, Yao Q, Wang J, Chen J, Eggleton SP, Liu T. Efficacy and Tolerability of First-Line Cetuximab Plus Leucovorin, Fluorouracil, and Oxaliplatin (FOLFOX-4) Versus FOLFOX-4 in Patients With RAS Wild-Type Metastatic Colorectal Cancer: The Open-Label, Randomized, Phase III TAILOR Trial. J Clin Oncol. 2018 Oct 20;36(30):3031-3039. doi: 10.1200/JCO.2018.78.3183. Epub 2018 Sep 10. PMID 30199311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to enroll subjects with Kirsten rat sarcoma viral oncogene homolog (KRAS) wild-type (wt) tumors.Following modification of approved EU indication of cetuximab,a decision made to amend study population from subjects with KRAS wt tumors to those with RAS wt tumors. All efficacy/safety analysis based on subjects with RAS wt tumor.
Pre-assignment Details: First subject first visit/last subject last visit: 30 September 2010/31 Jan 2018. A total of 553 subjects were enrolled in the trial. 504 subjects were randomized in the study, of which 397 were with RAS wt tumors. Participant Flow is presented for the subjects with RAS wt tumors.
Groups:
- Cetuximab + FOLFOX4: Subjects received cetuximab in combination with FOLFOX-4 chemotherapy regimen. FOLFOX-4 chemotherapy regimen consists of a combination of oxaliplatin with 5-fluorouracil (5-FU)/folinic acid (FA). Cetuximab was always administered every 7 days with an initial dose of 400 milligram per square meter (mg/m^2) at 5 milligram per minute (mg/min) and 250 mg/m^2 at 10 mg/min for subsequent infusions, followed by oxaliplatin 85 mg/m^2 infused over 120 minutes at least 1 hour later. Following completion of the oxaliplatin infusion or simultaneously with oxaliplatin, FA was administered at a dose of 200 mg/m^2 infused over 120 minutes, on Day 1, Day 2, and every 2 weeks and then 5- FU was administered as a bolus of 400 mg/m^2/day intravenously over 2-4 minutes followed by 600 mg/m^2/day infused over 22 hours, on Day 1, Day 2, and every 2 weeks. All subjects received treatment until progression of disease, withdrawal of consent, or unacceptable toxicity.
- FOLFOX4: Subjects received FOLFOX-4 chemotherapy regimen that consists of a combination of oxaliplatin with 5-FU/FA. Oxaliplatin 85 mg/m^2 infused over 120 minutes was administered first or simultaneously with FA at a dose of 200 mg/m^2 infused over 120 minutes on Day 1, Day 2, and every 2 weeks and then 5-FU was administered as a bolus of 400 mg/m^2/day intravenously over 2-4 minutes followed by 600 mg/m^2/day infused over 22 hours on Day 1, Day 2, and every 2 weeks. All subjects received treatment until progression of disease, withdrawal of consent, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cetuximab + FOLFOX4 | FOLFOX4
Started | 193 | 204
Modified Intent-to-treat Population | 193 | 200
Modified Safety Population | 194 (One subject was randomized to FOLFOX-4 group but received cetuximab + FOLFOX-4 treatment instead) | 199
Completed | 193 | 200
Not Completed | 0 | 4
Not completed — Randomized, but not treated | 0 | 4

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (MITT) population included all subjects with RAS wild-type tumor status who were randomized to study treatment and who received at least 1 dose of study treatment. Subjects were analyzed as randomized.
Groups:
- Cetuximab + FOLFOX-4: Subjects received cetuximab in combination with FOLFOX-4 chemotherapy regimen. FOLFOX-4 chemotherapy regimen consists of a combination of oxaliplatin with 5-FU/FA. Cetuximab was always administered every 7 days with an initial dose of 400 mg/m^2 at 5 mg/min and 250 mg/m^2 at 10 mg/min for subsequent infusions, followed by oxaliplatin 85 mg/m^2 infused over 120 minutes at least 1 hour later. Following completion of the oxaliplatin infusion or simultaneously with oxaliplatin, FA was administered at a dose of 200 mg/m^2 infused over 120 minutes, on Day 1, Day 2, and every 2 weeks and then 5- FU was administered as a bolus of 400 mg/m^2/day intravenously over 2-4 minutes followed by 600 mg/m^2/day infused over 22 hours, on Day 1, Day 2, and every 2 weeks. All subjects received treatment until progression of disease, withdrawal of consent, or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4 | Total
Number analyzed (Participants) | 193 | 200 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.8) | 55.1 (11.2) | 54.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 61 | 127
  Male | 127 | 139 | 266

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Time
Description: PFS was defined as the duration (in months) from randomization until the first progressive disease (PD) observation as assessed by the Independent Review Committee (IRC) according to Response Evaluation Criteria for Solid Tumors (RECIST) version 1.0, or death due to any cause when death occurred within 90 days of randomization or the last tumor assessment, whichever was later. PD was defined as at least a 20% increase in the sum of longest diameter (LD) of the target lesions, taking as references the smallest sum LD since the treatment started (including baseline), or appearance of one or more new lesions, and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline up to 333 weeks
Population: MITT population included all subjects with RAS wild-type tumor status who were randomized to study treatment and who received at least 1 dose of study treatment. Subjects were analyzed as randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4
Number analyzed (Participants) | 193 | 200
months | 9.2 [8.8 to 10.9] | 7.4 [5.8 to 7.5]
Statistical Analysis 1: Comparison: Cetuximab + FOLFOX-4 vs FOLFOX-4; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.629, 95% CI 2-sided [0.498 to 0.794]

2. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as the time (in months) from randomization to death. For subjects who were still alive at the analysis data cut-off date or who lost to follow-up, survival was censored at the last recorded date that the subject was known to be alive.
Time Frame: Baseline up to 333 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4
Number analyzed (Participants) | 193 | 200
months | 20.8 [16.3 to 23.5] | 16.5 [14.8 to 19.5]

3. Secondary Outcome: Best Overall Response Rate (ORR)
Description: The Best ORR was defined as the percentage of subjects having achieved complete response (CR) or partial response (PR) according to RECIST version 1.0 as determined by the IRC. CR: defined as disappearance of all target and all non-target lesions and no new lesions. PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters, no progression of non-target lesions and no new lesions.
Time Frame: Baseline up to 333 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4
Number analyzed (Participants) | 193 | 200
percentage of subjects | 66.3 [59.2 to 72.9] | 40.5 [33.6 to 47.7]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as time from randomization to date of the first occurrence of radiologically confirmed PD as determined by IRC, Clinical PD according to the Investigator's assessment (if radiological confirmation of PD by IRC was unavailable), discontinuation of treatment due to progression or adverse event, start of new anticancer therapy, withdrawal of consent, or death within 90 days of last tumor assessment or randomization. Subjects without event were censored on the date of last tumor assessment.
Time Frame: Baseline up to 333 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4
Number analyzed (Participants) | 193 | 200
months | 9.2 [7.4 to 9.3] | 5.6 [5.6 to 6.5]

5. Secondary Outcome: Number of Subjects With Curative Surgery of Liver Metastases
Description: The number of subjects who underwent liver metastatic surgery after start of treatment and the outcome of surgery with respect to residual tumor after surgery (R0, R1, R2, not evaluable) were summarized. In case of resection of more than one metastasis, the worst outcome of surgery defined the overall status of a subject. R0 = No residual tumor after resection (all lesions resected completely); R1 = Metastases not resected completely with microscopic residual lesions; and R2 = Metastases not resected completely with macroscopic residual lesions.
Time Frame: Baseline up to 333 weeks
Population: MITT population included all subjects with RAS wild-type tumor status who were randomized to study treatment and who received at least 1 dose of study treatment. Subjects were analyzed as randomized. Here "Number Analyzed" signifies those subjects who were evaluable for the specified categories.
Measure: Number; unit: subjects
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4
Number analyzed (Participants) | 193 | 200
subjects
  Subjects with liver surgery | 9 | 6
  Subjects with liver surgery outcome: R0 | 7 | 2
  Subjects with liver surgery outcome: R1 | 1 | 2
  Subjects with liver surgery outcome: R2 | 0 | 0
  Subjects not evaluable | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Safety Follow up (assessed up to 333 weeks)
Description: Modified safety population included all subjects with RAS wild type tumor status who received any study treatment (cetuximab, oxaliplatin or 5-FU/FA). Subjects were analyzed as treated.
Arm/Group | Cetuximab + FOLFOX-4 | FOLFOX-4
All-Cause Mortality (participants affected / at risk) | 157/194 | 173/199
Serious Adverse Events (participants affected / at risk) | 42/194 | 27/199
Other Adverse Events (participants affected / at risk) | 194/194 | 194/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + FOLFOX-4 (N=194) | FOLFOX-4 (N=199)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 2
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ANAL FISTULA (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
ENTERITIS (Gastrointestinal disorders) | 1 | 0
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 7 | 4
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 3 | 3
PYREXIA (General disorders) | 0 | 1
SUDDEN DEATH (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 2 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 1
ANAL ABSCESS (Infections and infestations) | 0 | 1
EPIDIDYMITIS (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 2
HEADACHE (Nervous system disorders) | 0 | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
URETERIC OBSTRUCTION (Renal and urinary disorders) | 2 | 0
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 2 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0
PHLEBITIS (Vascular disorders) | 0 | 2
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS LIMB (Vascular disorders) | 2 | 1
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 | 0
INFUSION SITE INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + FOLFOX-4 (N=194) | FOLFOX-4 (N=199)
ANAEMIA (Blood and lymphatic system disorders) | 28 | 24
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 18 | 14
LEUKOPENIA (Blood and lymphatic system disorders) | 151 | 146
NEUTROPENIA (Blood and lymphatic system disorders) | 156 | 149
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 92 | 102
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 21 | 13
ABDOMINAL PAIN (Gastrointestinal disorders) | 37 | 19
CONSTIPATION (Gastrointestinal disorders) | 43 | 29
DIARRHOEA (Gastrointestinal disorders) | 69 | 35
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 12 | 5
HAEMATOCHEZIA (Gastrointestinal disorders) | 10 | 5
MOUTH ULCERATION (Gastrointestinal disorders) | 22 | 9
NAUSEA (Gastrointestinal disorders) | 70 | 92
STOMATITIS (Gastrointestinal disorders) | 32 | 14
VOMITING (Gastrointestinal disorders) | 43 | 52
FATIGUE (General disorders) | 77 | 56
PYREXIA (General disorders) | 59 | 48
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 19 | 21
LIVER INJURY (Hepatobiliary disorders) | 12 | 6
DRUG HYPERSENSITIVITY (Immune system disorders) | 18 | 15
NASOPHARYNGITIS (Infections and infestations) | 10 | 4
PARONYCHIA (Infections and infestations) | 28 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 14
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 20 | 12
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 65 | 54
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 58 | 58
BLOOD ALBUMIN DECREASED (Investigations) | 12 | 4
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 16 | 8
BLOOD BILIRUBIN INCREASED (Investigations) | 15 | 7
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 11 | 11
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 12 | 11
HAEMOGLOBIN DECREASED (Investigations) | 28 | 42
NEUTROPHIL COUNT DECREASED (Investigations) | 11 | 13
PLATELET COUNT DECREASED (Investigations) | 19 | 18
WEIGHT DECREASED (Investigations) | 51 | 26
WEIGHT INCREASED (Investigations) | 23 | 14
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 14 | 9
DECREASED APPETITE (Metabolism and nutrition disorders) | 75 | 60
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 10 | 5
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 13 | 13
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 23 | 14
HYPONATRAEMIA (Metabolism and nutrition disorders) | 16 | 18
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 12 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 | 11
HYPOAESTHESIA (Nervous system disorders) | 25 | 27
NEUROTOXICITY (Nervous system disorders) | 15 | 18
INSOMNIA (Psychiatric disorders) | 11 | 10
INSOMNIA (Psychiatric disorders) | 10 | 10
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 | 16
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 31 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 17 | 7
PRURITUS (Skin and subcutaneous tissue disorders) | 10 | 3
RASH (Skin and subcutaneous tissue disorders) | 120 | 7
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 17 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 65 | 38
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 39 | 6
ASTHENIA (General disorders) | 11 | 13
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 7 | 11
DRY SKIN (Skin and subcutaneous tissue disorders) | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other